CLINICAL TRIAL: NCT06028815
Title: Effects of Group Music Therapy Intervention for Informal Caregivers of Elderly Dependents
Brief Title: Group Music Therapy Intervention With Informal Carers of Elderly Dependents
Acronym: MUSIC CARES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Deusto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NeuroemotionMusicCares
Record Dates: First submitted 2023-07-26; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Care Burden; Anxiety; Depression; Coping Strategies; Quality of Life
Keywords: Group music therapy; Informal caregivers; Health-related quality of life (HRQOL); Anxiety; Depression
MeSH Terms: conditions — Caregiver Burden; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Informal carers receive 10 music therapy sessions
  Interventions: Behavioral: Group music therapy
- Control group (No Intervention): Informal carers do not receive music therapy sessions

INTERVENTIONS:
Behavioral: Group music therapy — Music therapy intervention using active and receptive techniques, focusing on the technique of songwriting.
  Arms: Experimental group

SUMMARY:
To evaluate the effects of a group music therapy intervention with informal caregivers of elderly people on clinical psychological symptoms, taking into account variables such as caregiver burden, anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* to be the main informal caregiver of an elderly dependant
* the dependant person has to be over 60 years of age
* to be over 18 years of age
* having signed the informed consent form accepting the assessment and intervention

Exclusion Criteria:

* not residing in Spain
* being under 18 years
* having uncompensated sensory deficits that prevented the administration of the assessment protocol;
* illiteracy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-31 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life | 3 months
  For evaluating Health-Related Quality of Life is going to use the 36-Item Short Form Health Survey questionnaire (SF-36).
  The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). Component analyses showed that there are two distinct concepts measured by the SF-36: a physical dimension, represented by the Physical Component Summary (PCS), and a mental dimension, represented by the Mental Component Summary (MCS).
  The correct calculation of SF-36 summary measures PCS and MCS requires the use of special algorithms.
  The scores obtained in this questionnaire range from 0 to 100, with 0 being the worst state of health and 100 the best state of health for the dimension assessed. Thus, the higher the score obtained, the better the quality of life of the person assessed.
Anxiety Stay and Trait | 3 months
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety that also is often used in research as an indicator of caregiver distress.
  It has 20 items for assessing trait anxiety and 20 for state anxiety, on a 4-point Likert scale.
  Scores range from 20 to 80, with higher scores correlating with greater anxiety
Depression | 3 months
  Assessed with the BDI-II that contains 21 items and identifies symptoms and attitudes associated with depression.
  Each item is evaluated on a severity scale ranging from 0-3, with a total score ranging from 0-63.
  Higher total scores indicate more severe depressive symptoms
Burden | 3 months
  To assess the burden, it is using the Burden Zarit Interview that is a self-report instrument that assesses the level of caregiver burden. It consists of 22 items that are assessed using a Likert-type scale, where higher scores indicate greater burnout.

SECONDARY OUTCOMES:
Coping strategies | 3 months
  Coping strategies are evaluated with the COPE-28 that is the brief version inventory of 28 items and 14 subscales that is applied on an ordinal Likert-type scale with four response alternatives (from 0 to 3) between "I never do this" and "I always do this", with intermediate scores.
Spirituality | 3 months
  The outcome spirituality is assessed with the WHOQOL-SRPB,a 32-item instrument that measures spiritual, religious, and personal beliefs in 8 dimensions. Each item has a 5-point Likert format for responses from 1 ("not at all") to 5 ("completely").
  The WHOQOL-SRPB total score ranges from 0 to 100, with higher scores indicating higher spirituality.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Deusto, Bilbao, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data is available from now until 2025